CLINICAL TRIAL: NCT03786653
Title: Feasibility of Immunotherapy Administration to Patients With Bronchial Cancer in a Hospital-at- Home Setting - ImHADom
Brief Title: Feasibility of Immunotherapy Administration to Patients With Bronchial Cancer in a Hospital-at- Home Setting (ImHADom)
Acronym: ImHADom
Status: Completed | Type: Observational
Sponsor: RENAULT Patrick Aldo (Other)
Responsible Party: Sponsor-Investigator, RENAULT Patrick Aldo, Principal Investigator, Centre Hospitalier de PAU
Organization: Centre Hospitalier de PAU (Other)
Other Study IDs: CHPAU2018/02
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2021-01

CONDITIONS: Bronchial Cancer
Keywords: Immunotherapy, bronchial cancer, home-based hospitalization
MeSH Terms: conditions — Carcinoma, Bronchogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational prospective monosite study aims to describe, for the first time, management in a hospital-at-home programme of patients treated by immunotherapy for bronchial cancer.

The feasibility in good conditions of this management, the patients' quality of life and their satisfaction will be evaluated.

DETAILED DESCRIPTION:
Those last years, immunotherapy treatment for bronchial cancers allowed considerable progress in terms of tumoral answer, survival without progression and global survival. Usually administered in the day hospitalization department, its preparation and administration to the patient are compatible with hospital-at-home management. Currently, this offer of care is rarely proposed, and only in particular situations. At the Hospital of Pau, it was introduced recently. It is proposed to patients who have been receiving immunotherapy for at least 4 months. At the moment, there is no study stating the feasibility of home hospitalization for patients treated by immunotherapy. Given that there is neither regulatory obstacle nor any contraindication to care in home hospitalization, the choice of a descriptive study stands out.

This study will be proposed to all the patients for whom home hospitalization has been decided and scheduled by the healthcare team in a medical staff meeting.

The patients included in the study will be followed according to the common practice: a consultation every 3 months during 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over.
* with bronchial cancer treated with immunotherapy,
* having two assessments of the response to immunotherapy received in day hospitalization with efficiency (stability or partial response)
* without any graded higher than 1 adverse effects, or uncontrolled grade 1 adverse effects related to immunotherapy
* eligible for a home-based hospitalization

Exclusion Criteria:

* Patient receiving immunotherapy via temporary authorization for use,
* Frail patients requiring a frequent medical assessment thus day hospitalization cares

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by immunotherapy for bronchial cancer
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of home-based immunotherapy (percentage of patients who interrupted their home hospitalization for reasons directly linked to that management) | 1 year
  Feasibility under good conditions of home-based immunotherapy, defined by the percentage of patients who interrupted their home hospitalization for reasons directly linked to that management.

SECONDARY OUTCOMES:
adverse effects | 1 year
  Immunotherapy related adverse effects monitoring criteria evaluation
Number of Incidents occurring during the Hospital at Home program handling process | 1 year
  The occurrence of possible incidents related to the Hospital at Home program will be collected at each home based hospitalization.
Quality of Life Questionnaire (EORTC QLQ-C30) total score | at inclusion, month 3, 6 9 and 12
  To study the patient's reported quality of life before and throughout therapy. Quality of life score obtained through self-administered EORCT QLQ-C30 questionnaire at inclusion, month 3, 6 9 and 12.
Patients' Satisfaction Questionnaire | 1 year
  Patients' satisfaction with their home base management will be assessed with a questionnaire. It will be collected at month 3, 6 9 and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier de pau, Pau, Aquitaine, France